CLINICAL TRIAL: NCT05651607
Title: Evaluation of the Efficacy of CANNABIDIOL on the Pruritus in Children With Hereditary Epidermolysis Bullosa
Acronym: EBCBD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: HELEBOR (Unknown); Fondation Apicil (Other); Lions Club International Foundation (Other); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP220741; 2022-003411-28 (EudraCT Number)
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2023-09

CONDITIONS: Hereditary Epidermolysis Bullosa
Keywords: hereditary epidermolysis bullosa; Cannabidiol; Prutitus; Pilot Study
MeSH Terms: interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cannabidiol (Epidyolex) (Experimental)
  Interventions: Drug: Cannabidiol

INTERVENTIONS:
Drug: Cannabidiol — Oral solution, taken 3 times a day (morning, noon and evening), 5 mg/kg/day from day D0 to day D4. If not effective and well tolerated, dose increase : 10 mg/kg/day from day D5 to day D9, then 20 mg/kg/day from day D10 to day D29, maximum 800 mg/day
  Other Names: Epidyolex

SUMMARY:
Hereditary epidermolysis bullosa (HEB) is a heterogeneous group of rare genetic diseases, characterized by fragility of the skin and mucous membranes, which results in the appearance of mucocutaneous bullae and erosions during minimal trauma. Pruritus is a neuropathic pain mainly related to activation of unmyelinated cutaneous C nerve fibers and is very common in patients with HEB. It is the cause of trophic disorders, aggravation of certain wounds, appearance of new bubbles. In addition, this chronic pruritus can also have a major psychological impact on the patient and his family. However, these therapies used in the pruritus of patients with HEB have often proven to be ineffective.

In order to improve the quality of life of children and their families, research into new therapies to limit this chronic pruritus is necessary. Among phytocannabinoids, CANNABIDIOL (CBD) should be clearly distinguished from Delta-9-tetrahydrocannabinol (THC). Indeed, CBD is an "inverse" agonist of the CB2 receptor, it acts by reducing the effect of this receptor, while THC is an agonist of the CB1 and CB2 receptors. Thus, CBD has antipsychotic, anxiolytic, antiemetic, anti-inflammatory and anti-epileptic effects, unlike THC which has psychotic, relaxation effects, impairs cognitive function and memory. Cannabinoids are involved in the physiopathology in pruritus at the level of the peripheral nervous system via the CB1 and TRPV1 receptors, and also at the level of the central nervous system thanks to the CB1 and CB2 receptors. In addition, inflammation plays an important role in the physiopathology of pruritus and this is reduced via the activation of CB2 receptors, expressed in immune cells. Various studies with promising results have examined the effect of cannabinoids in pruritus. No serious adverse effects have been reported and the rare adverse effects that have been observed are reversible upon discontinuation of treatment.

The research project seeks to estimate the efficacy of CANNABIDIOL in the pruritus of 10 children with severe hereditary epidermolysis bullosa. Pruritus is assessed before the start of treatment, then after one month of taking oral treatment, three times a day. The effectiveness of taking the treatment will also be assessed on pain, on the impact on sleep and on overall quality of life. The tolerance of CANNABIDIOL will be well monitored. The systemic passage of CANNABIDIOL is measured during a routine blood test 1 month after treatment.

DETAILED DESCRIPTION:
Experimental scheme M-3 to M-1: pre-inclusion Proposal of the study and information of the families followed in the dermatology department during a visit as part of the care pathway. Explanation of protocol.

D0: inclusion

During conventional hospitalization or day hospitalization of the patient in the dermatology department for monitoring of hereditary epidermolysis bullosa (EBH) :

* Signature of the consent of the legal guardians after verification of the eligibility criteria and information given on the protocol
* Collection of pruritus and pain scores
* Clinical skin examination with measurement of the severity score of epidermolysis bullosa EBDASI (Epidermolysis Bullosa Disease Activity and Scarring Index).
* List of treatments and medical devices of the patient
* Quality of sleep measured by the patient or his family on a scale of 0 to 10
* Quality of life measured by the patient or his family via the child DLQI questionnaire

  1. st intake of CANNABIDIOL D0 to D4: 5 mg/kg/day in 3 doses (morning, noon and evening). on D5: If efficacy (mean VAS for pruritus <3 on D4), continue at the same dosage. If ineffective or partially effective (VAS pruritus ≥3) and in the event of good tolerance, increase to 10 mg/kg/day in 3 doses (morning, noon and evening).

on D10: If efficacy (mean VAS pruritus <3 on D9), continue at the same dosage. If ineffective or partially effective (VAS pruritus ≥3), and in the event of good tolerance, increase to 20 mg/kg/day in 3 doses (morning, noon and evening) if previous dosage at 10 mg/kg/day, or increase to 10 mg/kg/day if previous dosage at 5 mg/kg/day.

In case of intolerance at D5, D10, D14 or D21: decrease to the previous dosage, or interruption if the dosage was 5 mg/kg/day.

D30(+/-2): end of treatment consultation The end-of-treatment consultation takes place D30 (+/-2) after the start of treatment.

* Collection of pruritus and pain scores
* Clinical skin examination with measurement of the EBDASI score
* Quality of sleep measured by the patient or his family on a scale of 0 to 10
* Quality of life measured by the patient or his family via the child DLQI questionnaire
* During a systematic blood test, collection of two more tubes for CANNABIDIOL dosage and a liver test

D48 (+2): phone call by the investigating doctor to monitor the occurrence of adverse events

ELIGIBILITY:
Inclusion Criteria:

* Minor patient between 2 and 17 years and 10 months
* Suffering from distrophic recessive epidermolysis bullosa
* Patient weight less than or equal to 40 kg
* With pruritus not relieved by conventional treatments with mean VAS greater than or equal to 4/10 the 3 days preceding inclusion
* No change in treatment or care for at least one month
* Consent of parents
* Affiliated to social security

Exclusion Criteria:

* Hypersensitivity to the active substance or to any of the excipients (Refined sesame oil, anhydrous ethanol, sucralose, strawberry flavor, includes benzyl alcohol)
* Consumption of cannabis or cannabidiol
* Severe renal impairment defined by GFR less than 29 ml/min
* Moderate to severe hepatic impairment defined by a Child-Pugh B or C score or an AST and/or ALT level greater than 3 times normal and/or bilirubin more than 2 times normal
* with clinically or ultrasound sign(s) of moderate to severe cardiac insufficiency, defined by LVEF less than 45% and stage II to IV of the NYHA classification
* Taking a tricyclic antidepressant treatment with anti-H4 antihistamine action or a neurokinin-1 receptor antagonist in the previous month
* Participating to an interventional research (category 1 or 2)
* Modification of at least one background treatment in the previous month
* Proven pregnancy or breastfeeding patient
* Patient deprived of their liberty by decision of a judicial or administrative authority (Article L. 1121-6 of the Public Health Code)

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2023-09-07 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Clinically significant decrease of pruritus Visual Analog Scale (VAS) scores | Day 30
  Loss of at least 2 points on the mean pruritus VAS scores recorded on D27, D28 and D29 compared to the mean pruritus scores recorded on D-3, D-2 and D-1 (D0 = inclusion and start of treatment). The Visual Analogue Scale (VAS) is a scale consisting of a 10cm long line and a single question. The scale is scored in a range of 0-10 with 10 representing worst imaginable pruritus.

SECONDARY OUTCOMES:
Change of pruritus Visual Analog Scale scores | Day 30
  Change of the mean pruritus VAS scores recorded on D27, D28 and D29 compared to the mean pruritus VAS scores on D-3, D-2 and D-1 . The scale is scored in a range of 0-10 with 10 representing worst imaginable pruritus.
Evaluation of tolerance of Cannabidiol | Day 48
  Serious and non-serious side effects
Clinically significant decrease of chronic pain scores | Day 30
  Loss of at least 2 points on the mean pain scores (VAS or FLACC according to the age of patient) recorded on D27, D28 and D29 compared to the mean pain scores recorded on D-3, D-2 and D-1 (D0 = inclusion and start of treatment). The Face, Legs, Activity, Cry, Consolability (FLACC) scale is a measurement used to assess pain for children between the ages of 2 months and 7 years or individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 10 representing severe pain.
  The Visual Analogue Scale (VAS) is a scale consisting of a 10cm long line and a single question. The scale is scored in a range of 0-10 with 10 representing worst imaginable pain.
Change of chronic pain scores | Day 30
  Change of the mean pain scores (Visual Analogue Scale or Face, Legs, Activity, Cry, Consolability scale according to the age of patient) recorded on D27, D28 and D29 compared to the mean pain scores on D-3, D-2 and D-1 The Face, Legs, Activity, Cry, Consolability (FLACC) scale is a measurement used to assess pain for children between the ages of 2 months and 7 years or individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 10 representing severe pain.
  The Visual Analogue Scale (VAS) is a scale consisting of a 10cm long line and a single question. The scale is scored in a range of 0-10 with 10 representing worst imaginable pain.
Change of pruritus Visual Analog Scale score during cares | Day 30
  Change of the mean of maximum pruritus VAS scores recorded during the last two cares before D30 compared to the mean of maximum pruritus VAS scores recorded during the last two cares before D0. The Visual Analogue Scale (VAS) is a scale consisting of a 10cm long line and a single question. The scale is scored in a range of 0-10 with 10 representing worst imaginable pruritus.
Change of acute pain score during cares | Day 30
  Change of the mean of maximum acute pain scores (VAS or FLACC according to the age of patient) recorded during the last two cares before D30 compared to the mean of maximum acute pain scores recorded during the last two cares before D0. The Face, Legs, Activity, Cry, Consolability (FLACC) scale is a measurement used to assess pain for children between the ages of 2 months and 7 years or individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 10 representing severe pain.
  The Visual Analogue Scale (VAS) is a scale consisting of a 10cm long line and a single question. The scale is scored in a range of 0-10 with 10 representing worst imaginable pain.
Change of quality of sleep | Day 30
  Quality of sleep measured by the patient or his family on a scale of 0 to 10, with 10 representing excellent sleep quality, at D30 compared to D0
Change of quality of life | Day 30
  Quality of life measured by the patient or his family via the Dermatology Life Quality Index (DLQI child) at D30 compared to D0.
  The Dermatology Life Quality Index (DLQI child) is scored in a range of 0-30 with 30 representing extremely important effect on the patient's quality life.
Systemic passage of CANNABIDIOL | Day 30
  Systemic passage measured at D30 by blood test 4 hours after the morning intake and before the midday intake of CANNABIDIOL.
Acceptability of CANNABIDIOL | Day 30
  Measure of acceptability: difficulty of ingesting, difficulty of using the syringe, taste

CONTACTS AND LOCATIONS:
Overall Officials: Christine BODEMER, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris; Lara MAYRAND, Resident, Study Chair — Assistance Publique - Hôpitaux de Paris; Céline GRECO, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sivesind TE, Maghfour J, Rietcheck H, Kamel K, Malik AS, Dellavalle RP. Cannabinoids for the Treatment of Dermatologic Conditions. JID Innov. 2022 Jan 13;2(2):100095. doi: 10.1016/j.xjidi.2022.100095. eCollection 2022 Mar. PMID 35199092
- [Background] Sheriff T, Lin MJ, Dubin D, Khorasani H. The potential role of cannabinoids in dermatology. J Dermatolog Treat. 2020 Dec;31(8):839-845. doi: 10.1080/09546634.2019.1675854. Epub 2019 Oct 10. PMID 31599175
- [Background] Eagleston LRM, Kalani NK, Patel RR, Flaten HK, Dunnick CA, Dellavalle RP. Cannabinoids in dermatology: a scoping review. Dermatol Online J. 2018 Jun 15;24(6):13030/qt7pn8c0sb. PMID 30142706
- [Background] Avila C, Massick S, Kaffenberger BH, Kwatra SG, Bechtel M. Cannabinoids for the treatment of chronic pruritus: A review. J Am Acad Dermatol. 2020 May;82(5):1205-1212. doi: 10.1016/j.jaad.2020.01.036. Epub 2020 Jan 25. PMID 31987788
- [Background] Stander S, Reinhardt HW, Luger TA. [Topical cannabinoid agonists. An effective new possibility for treating chronic pruritus]. Hautarzt. 2006 Sep;57(9):801-7. doi: 10.1007/s00105-006-1180-1. German. PMID 16874533
- [Background] Okusanya BO, Asaolu IO, Ehiri JE, Kimaru LJ, Okechukwu A, Rosales C. Medical cannabis for the reduction of opioid dosage in the treatment of non-cancer chronic pain: a systematic review. Syst Rev. 2020 Jul 28;9(1):167. doi: 10.1186/s13643-020-01425-3. PMID 32723354
- [Background] Schrader NHB, Gorell ES, Stewart RE, Duipmans JC, Harris N, Perez VA, Tang JY, Wolff AP, Bolling MC. Cannabinoid use and effects in patients with epidermolysis bullosa: an international cross-sectional survey study. Orphanet J Rare Dis. 2021 Sep 6;16(1):377. doi: 10.1186/s13023-021-02010-0. PMID 34488820
- [Background] Chelliah MP, Zinn Z, Khuu P, Teng JMC. Self-initiated use of topical cannabidiol oil for epidermolysis bullosa. Pediatr Dermatol. 2018 Jul;35(4):e224-e227. doi: 10.1111/pde.13545. Epub 2018 May 22. PMID 29786144
- [Background] Schrader NHB, Duipmans JC, Molenbuur B, Wolff AP, Jonkman MF. Combined tetrahydrocannabinol and cannabidiol to treat pain in epidermolysis bullosa: a report of three cases. Br J Dermatol. 2019 Apr;180(4):922-924. doi: 10.1111/bjd.17341. Epub 2018 Nov 14. PMID 30347109
- [Background] Welponer T, Diem A, Nahler G, Laimer M. Purified oral cannabidiol for pain management in severe recessive dystrophic epidermolysis bullosa. Indian J Dermatol Venereol Leprol. 2022 May-Jun;88(4):551-552. doi: 10.25259/IJDVL_71_2021. No abstract available. PMID 35593277